CLINICAL TRIAL: NCT00000918
Title: A Phase II, Randomized, Open-Label Comparative Trial of Salvage Antiretroviral Therapies for HIV-Infected Individuals With Virological Evidence of Nelfinavir Treatment Failure as Reflected by Plasma HIV RNA Concentration of >= 1,000 Copies/ml
Brief Title: A Study to Compare The Ability of Different Anti-HIV Drugs to Decrease Viral Load After Nelfinavir (an Anti-HIV Drug)Treatment Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 400; 11356 (Registry Identifier: DAIDS ES Registry Number); Substudy A5013s; Substudy A5022s
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Reverse Transcriptase Inhibitors; Salvage Therapy; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; lamivudine, zidovudine drug combination; Ritonavir; amprenavir; efavirenz; Saquinavir; Lamivudine; Stavudine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine/Zidovudine
Drug: Ritonavir
Drug: Amprenavir
Drug: Efavirenz
Drug: Saquinavir
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of combining several anti-HIV drugs in order to decrease plasma viral load (level of HIV in the blood) in HIV-positive patients who have failed nelfinavir (NFV) treatment.

In order to determine the ability of a drug regimen to decrease viral load after drug treatment has failed, it is best to test a variety different of drug "cocktails" (drug regimens). The drug cocktails in this study include 2 new nucleoside reverse transcriptase inhibitors (NRTIs), efavirenz (an NNRTI, non-nucleoside reverse transcriptase inhibitor), and either 1 or 2 protease inhibitors. It is important to include multiple drugs from different groups in a drug cocktail since combinations containing fewer drugs are likely to fail.

DETAILED DESCRIPTION:
To maximize the likelihood of a favorable response to salvage therapy, 4 or 5 drug regimens should be studied. Regimens containing fewer drugs, particularly those lacking a non-nucleoside reverse transcriptase inhibitor (NNRTI) such as efavirenz, are likely to result in an unacceptable rate of virological failure. Therefore, this study examines drug combinations which include two new nucleoside reverse transcriptase inhibitors (NRTIs), the NNRTI efavirenz, and either one or two protease inhibitors which are known not to produce cross-resistance to nelfinavir.

Patients are randomly selected to receive 1 of the following 4 treatment regimens:

Arm A: Ritonavir, saquinavir, efavirenz, and 2 new NRTIs. Arm B: Indinavir, efavirenz and 2 new NRTIs. Arm C: Amprenavir, efavirenz, and 2 new NRTIs. [AS PER AMENDMENT 3/22/00: Patients have the option to increase the APV dose or to add low-dose ritonavir. APV will continue to be provided by the study; ritonavir will not be provided by the study.] Arm D: Indinavir, amprenavir, efavirenz, and 2 new NRTIs. [AS PER AMENDMENT 6/28/99: All treatment regimens must include at least 1 new NRTI.] [AS PER AMENDMENT 3/22/00: ACTG 400 will continue to provide originally randomized study medications to all patients until approximately May 10, 2000, regardless of virologic response. Patients may also add antiretrovirals of their choice to this regimen (not provided by the study).] Clinical assessments are taken at Weeks 2, 4, 8, 12, 16, and every 8 weeks thereafter for the duration of the study. In addition, 2 substudies are being conducted: a drug-interaction substudy and a drug-exposure substudy. [AS PER AMENDMENT 3/22/00: Both substudies are closed to accrual and their pharmacokinetics assessments are discontinued.]

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are over 13 years old (need consent of parent or guardian if under 18).
* Are HIV-positive.
* Currently have virologic failure (more than 1,000 copies of HIV RNA per ml).
* Agree to abstinence or use of effective birth control during the study.
* Have been taking NFV for the past 12 weeks.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have a fever for 7 days or diarrhea for 30 days before study entry.
* Have a history of peripheral neuropathy within 60 days of study entry.
* Have hepatitis.
* Have any malignancy (cancer) other than minimal Kaposi's sarcoma.
* Are pregnant or breast-feeding.
* Are receiving radiation, chemotherapy, or any therapy for any illness within 14 days of study entry.
* Have taken amprenavir, saquinavir, indinavir or ritonavir for more than 7 days.
* Have received an HIV vaccine 30 days before study entry.
* Are receiving certain other medications.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Study Completion 2002-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mellors; William Powderly, Study Chair; Scott Hammer, Study Chair
Locations (39):
- United States (38):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Willow Clinic, Menlo Park, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - San Francisco Gen Hosp, San Francisco, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - Marin County Specialty Clinic, San Rafael, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Howard Univ, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Chelsea Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Washington, Seattle, Washington
- Univ of Puerto Rico, San Juan, Puerto Rico